CLINICAL TRIAL: NCT02295020
Title: Effect of Bioskin Ten-7 vs. Standard Treatment on Patient Reported Outcomes and Cytokine.
Acronym: Bioskin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cropper Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8627
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Anti-Inflammatory Agents, Non-Steroidal; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment Only (Active Comparator): Group A will receive standard treatment only such as NSAIDs and injections
  Interventions: Drug: Standard treatment only
- Standard Treatment plus Bioskin Ten-7 (Experimental): Group B will receive standard treatment such as NSAIDs and injections and the Bioskin Ten-7 knee brace.
  Interventions: Drug: Standard treatment only; Device: Standard treatment plus Bioskin Ten-7 knee brace

INTERVENTIONS:
Drug: Standard treatment only — Standard treatment such as NSAIDs and injections
  Other Names: NSAIDs and injections
Device: Standard treatment plus Bioskin Ten-7 knee brace — Standard treatment such as NSAIDs and injections plus Bioskin Ten-7 knee brace.
  Arms: Standard Treatment plus Bioskin Ten-7

SUMMARY:
The objectives of the study are 1.) to evaluate pain relief following the application of the Bioskin Ten-7 knee brace and 2.) to determine if use of the Bioskin Ten-7 knee brace is more effective at reducing inflammation than standard of care alone using synovial fluid cytokine analysis and validated outcome measures.

DETAILED DESCRIPTION:
Once consented, the patient is assigned to either Group A or Group B. Group A patients will receive standard treatment only and will not be prescribed a knee brace. Group B patients will receive standard treatment and the Bioskin Ten-7 knee brace. On Day 0, the patient will be assigned to one of the 2 groups using a 1:1 assignment. VAS, WOMAC, Oxford Knee Score, KOOS questionnaires will be administered and a sample of the patient's synovial fluid will be sent to labs for cytokine and cell count analysis. All patients will record use of NSAIDs and for Group B, the start and end time of brace use will be recorded. All patients will return in 8 weeks to assess efficacy of treatment. All patients will return their diaries, complete the same validated outcome measures as Day 0 and undergo a repeat synovial fluid analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years and older with primary diagnosis of Knee OA with no other knee diagnosis.
* Must have telephone access.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Dasa, MD, Principal Investigator — LSUHSC-NO, Orthopaedic Department

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment Only.: Group A will receive standard treatment only
  Standard treatment: Standard treatment such as NSAIDs and injections
- Standard Treatment Plus Bioskin Ten-7.: Group B will receive standard treatment and the Bioskin Ten-7 knee brace.
  Standard treatment: Standard treatment such as NSAIDs and injections
  Standard treatment plus Bioskin Ten-7 knee brace: Standard treatment such as NSAIDs and injections plus knee brace
Period: Overall Study
Arm/Group | Standard Treatment Only. | Standard Treatment Plus Bioskin Ten-7.
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment Only: Standard treatment only such as NSAIDs and injections
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.3) | 61.5 (8.8) | 59.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Standard of care [Number; unit: participants]
  Surpatz | 2 | 0 | 2
  NSAID | 14 | 4 | 18
  Medications | 4 | 16 | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (5.8) | 30.4 (4.3) | 32.4 (5.4)
KOOS - Pain [Mean (Standard Deviation); unit: units on a scale] — KOOS = Knee injury and Osteoarthritis Outcome Score. Pain refers to the pain sub-score.The scale is 0 to 100 where 100 indicates no problems and 0 indicates extreme problems.
  units on a scale | 37.8 (18.7) | 33.5 (20.3) | 35.6 (19.4)
KOOS - Symptoms [Mean (Standard Deviation); unit: units on a scale] — KOOS = Knee injury and Osteoarthritis Outcome Score. Symptoms refers to the Symptoms sub-score.The scale is 0 to 100 where 100 indicates no problems and 0 indicates extreme problems.
  units on a scale | 45.5 (22.4) | 35.6 (16.7) | 40.4 (20.1)
KOOS - ADL [Mean (Standard Deviation); unit: units on a scale] — KOOS = Knee injury and Osteoarthritis Outcome Score. ADL refers to the activities of daily living sub-score. The scale is 0 to 100 where 100 indicates no problems and 0 indicates extreme problems.
  units on a scale | 40.8 (15.6) | 37.2 (22.2) | 39.0 (19.1)
KOOS - Sport/Rec [Mean (Standard Deviation); unit: units on a scale] — KOOS = Knee injury and Osteoarthritis Outcome Score. Sport/Rec refers to the sport and recreational activities sub-score. The scale is 0 to 100 where 100 indicates no problems and 0 indicates extreme problems.
  units on a scale | 29.3 (25.9) | 12.1 (17.1) | 19.8 (22.9)
KOOS - QOL [Mean (Standard Deviation); unit: units on a scale] — KOOS = Knee injury and Osteoarthritis Outcome Score. QOL refers to the quality of life sub-score. The scale is 0 to 100 where 100 indicates no problems and 0 indicates extreme problems.
  units on a scale | 28.7 (19.6) | 14.4 (13.8) | 20.9 (18.0)
IL-6 [Median (Full Range); unit: pg/mL] | 1639 [49.9 to 25426] | 1309 [9.2 to 7905] | 1467.1 [9.2 to 25426]
IL-8 [Median (Full Range); unit: pg/mL] | 653.3 [19.2 to 4043] | 486.5 [8.9 to 7802] | 643.0 [8.9 to 7802]
TNF-alpha [Median (Full Range); unit: pg/mL] | 108.1 [7.7 to 1079] | 104.8 [2.1 to 436.8] | 108.1 [2.1 to 1079]
MIP-1alpha [Median (Full Range); unit: pg/mL] | 255.5 [1.2 to 24590] | 162.2 [4.2 to 2069] | 250.8 [1.2 to 24590]
MCP-1 [Median (Full Range); unit: pg/mL] | 8664 [1233 to 24831] | 10944 [876.7 to 21443] | 10188 [876.7 to 24831]

OUTCOME MEASURES:

1. Primary Outcome: KOOS - Pain
Description: Value at 8 weeks - value at day 0
Time Frame: Week 8- Day 0
Population: Discrepancies between participants flow chart and number of participants analyzed is due to patients not filling out the survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 16 | 17
units on a scale | 17.6 [8.4 to 26.8] | 9.1 [0.2 to 18.0]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.181, t-test, 2 sided

2. Primary Outcome: KOOS - Symptoms
Description: Value at 8 weeks - value at day 0
Time Frame: Week 8 - Day 0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment Only. | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 16 | 17
units on a scale | 10.6 [1.7 to 19.5] | 3.2 [-5.4 to 11.8]
Statistical Analysis 1: Comparison: Standard Treatment Only. vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.232, t-test, 2 sided

3. Primary Outcome: KOOS - ADL
Description: Value at 8 weeks - value at day 0
Time Frame: week 8 - day 0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 16 | 17
units on a scale | 15.3 [7.4 to 23.2] | 9.8 [2.1 to 17.4]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.311, t-test, 2 sided

4. Primary Outcome: KOOS - Sport/Rec
Description: Value at 8 weeks - value at day 0
Time Frame: Week 8 - day 0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 12 | 12
units on a scale | 13.8 [-3.5 to 31.0] | 9.6 [-7.6 to 26.8]

5. Primary Outcome: KOOS - QOL
Description: Value at 8 weeks - value at day 0
Time Frame: Week 8 - day 0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 14 | 16
pg/mL | 11.0 [0.2 to 21.8] | 5.4 [-4.7 to 15.6]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.449, t-test, 2 sided

6. Primary Outcome: Synovial Fluid Analysis (IL-6)
Description: Interleukine 6 in Synovial fluid analysis
Time Frame: Week 8 - day 0
Population: Discrepancies between participants flow chart and number of participants analyzed is due to either synovial fluid not present in the knee or not sufficient to be analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 10 | 11
pg/mL | -453.8 [-19670 to 18168] | -1055 [-7483 to 10399]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.860, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Synovial Fluid Analysis (IL-8)
Description: Interleukine 8 in Synovial fluid analysis
Time Frame: Week 8 - day 0
Population: as for outcome 6
Measure: Median (Full Range); unit: pg/mL
Groups:
- Standard Treatment Plus Bioskin Ten-7 Knee Brace: Standard treatment such as NSAIDs and injections plus knee Bioskin Ten-7 knee brace
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 11 | 12
pg/mL | -379.8 [-2875 to 6878] | -488.9 [-3542 to 4906]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.735, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Synovial Fluid Analysis (TNF-alpha)
Description: Tumor necrosis factor - alpha in Synovial fluid analysis
Time Frame: Week 8 - day 0
Population: as for outcome 6
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 11 | 12
pg/mL | -97.4 [-242.3 to 172.4] | -51.7 [-430.0 to 280.9]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.479, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Synovial Fluid Analysis (MIP - 1alpha)
Description: Macrophage Inflammatory Proteins - 1alpha
Time Frame: Week 8 - day 0
Population: as for outcome 6
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 9 | 11
pg/mL | -246.7 [-821.2 to 575.2] | -49.8 [-756.6 to 1715]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.323, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Synovial Fluid Analysis (MCP - 1)
Description: Monocyte chemotactic protein-1 - 1
Time Frame: Week 8 -day 0
Population: as for outcome 6
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Standard Treatment Only | Standard Treatment Plus Bioskin Ten-7 Knee Brace
Number analyzed (Participants) | 11 | 12
pg/mL | -7170 [-14933 to 17960] | -4890 [-15989 to 17432]
Statistical Analysis 1: Comparison: Standard Treatment Only vs Standard Treatment Plus Bioskin Ten-7 Knee Brace; Test type: Superiority or Other; p = 0.878, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Oxford Knee Score
Time Frame: Day 0 and Week 8
Population: The outcome was not measured as KOOS was measured as the only patient reported outcome.
Groups:
- Group A: Group A will receive standard treatment only
  Standard treatment: Standard treatment such as NSAIDs and injections
- Group B: Group B will receive standard treatment and the Bioskin Ten-7 knee brace.
  Standard treatment: Standard treatment such as NSAIDs and injections
  Standard treatment plus Bioskin Ten-7 knee brace: Standard treatment such as NSAIDs and injections plus knee brace
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: WOMAC
Description: assess pain, stiffness, and physical function measured by Western Ontario and McMaster universities Osteoarthritis Index
Time Frame: Day 0 and Week 8
Population: The outcome was not measured as KOOS was measured as the only patient reported outcome.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Visual Analog Scale
Description: identifies pain level
Time Frame: Day 0 and Week 8
Population: The outcome was not measured as KOOS was measured as the only patient reported outcome.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=20) | Group B (N=20)
CVA (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No